CLINICAL TRIAL: NCT07138196
Title: A Phase 1b, Open-label Dose Escalation Study to Evaluate the Safety, Pharmacodynamic, Pharmacokinetic and Preliminary Efficacy of Q702 in Subjects With Relapsed or Refractory Active Chronic Graft-versus-Host Disease (cGVHD)
Brief Title: A Study to Evaluate Adrixetinib (Q702) in Adults With Active Chronic Graft-Versus-Host Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QRNT-012
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Graft-Versus-Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adrixetinib (Q702) (Experimental): Escalating doses of adrixetinib in 28 day cycles.
  Interventions: Drug: Adrixetinib

INTERVENTIONS:
Drug: Adrixetinib — Administered orally
  Other Names: Q702

SUMMARY:
Open-label, dose escalation study to evaluate safety, tolerability pharmacokinetic and pharmacodynamic activity, and efficacy of Adrixetinib (Q702) in subjects with relapsed or refractory active chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are allogeneic HSCT recipients with moderate or severe active cGVHD requiring systemic immune suppression.
2. Subjects with relapsed or refractory active cGVHD who have progressed after all available standard of care treatments.
3. Subject must have documented progressive disease as defined by the NIH 2014 consensus criteria, in terms of either organ specific algorithm or global assessment, or active, symptomatic cGVHD for which the treating physician believes that a new line of systemic therapy is required.
4. Adequate organ and bone marrow functions.
5. Karnofsky Performance Scale of ≥ 60.

Exclusion Criteria:

1. Exposure to CSF1R inhibitor therapy for any indication after allogeneic transplant.
2. Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer.
3. Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years of enrollment.
4. Female subject who is pregnant or breastfeeding.
5. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2029-10-23 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLTs) | Cycle 1 (28 Days)
  DLTs assessed for each dose level
Number of Participants with Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs) | Cycle 1 (28 Days)
  AEs and SAEs assessed for each dose level.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Estimated up to Cycle 1 (28 Days)
  Maximum Observed Plasma Concentration (Cmax), area under the curve AUC of Q702 and its primary metabolites

OTHER OUTCOMES:
Objective Response Rate (ORR) | Cycle 7 Day 1 (One Cycle is 28 Days)
  Proportion of subjects with CR or PR by Cycle 7 Day 1 using Organ-specific response rate based on 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD
Duration of Response (DOR) | First CR or PR until documented PD, start of new therapy or death (Estimated up to 24 months)
  DOR defined as the time from best response of PR or CR until documented progression of cGVHD, start of new therapy, or death for any reason
Failure-Free Survival (FFS) | Baseline to, whichever occurs first of, PD, Addition of Systemic Immune Suppressive Therapy, or Death due to Any Cause (Estimated up to 24 months)
  FFS is defined as the time from study enrollment (first date of Q702 treatment) to addition of another systemic therapy for cGVHD, relapse of underlying malignancy, or death whichever is earlier.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto de Investigacion Sanitaria, Valencia

IPD SHARING:
Plan to Share IPD: Undecided